CLINICAL TRIAL: NCT01314547
Title: Impact of Environmental Factors on Disease Activity in Spondyloarthritis (SPA): Results of the Prospective Co-Env Cohort
Acronym: CoEnv
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AOM02020
Record Dates: First submitted 2011-03-11; First posted 2011-03-14 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2010-11

CONDITIONS: Spondylarthritis; Primary Systemic Vasculitis
Keywords: Environment; spondylarthritis; vasculitis; stress; life event; vaccine
MeSH Terms: conditions — Spondylarthritis; Vasculitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Susceptibility to SPA has been shown to be largely genetically determined. The objective of this study was to prospectively investigate the impact of several environmental factors on disease activity.

DETAILED DESCRIPTION:
Susceptibility to SPA has been shown to be largely genetically determined but the contribution of environmental factors to disease evolution has not yet been elucidated. The objective of this study was to prospectively investigate the impact of several environmental factors on disease activity.

ELIGIBILITY:
Inclusion Criteria:

* 18 years SPONDILARTHRITIS: modified New York criteria Systemic vasculitis: ACR criteria

Exclusion Criteria:

no internet access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with SPA disease
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2005-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Score on a disease activity rating scale | Six years
  Score on a disease activity rating scale (quaterly,than monthly basis)

SECONDARY OUTCOMES:
Ancillary studies will be possible with the available database | six years
  Ancillary studies will be possible with the available database

CONTACTS AND LOCATIONS:
Overall Officials: THOMAS HANSLIK, PU-PH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- hopital ambroise Pare, Boulogne, France